CLINICAL TRIAL: NCT00628693
Title: Quantitative Measurement of Cardiopulmonary Resuscitation During In Hospital Cardiac Arrest
Brief Title: Quantitative Measurement of Cardiopulmonary Resuscitation (CPR) During In Hospital Cardiac Arrest
Acronym: Q-CPR
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-6-4839; 1K23HD062629-01A1 (NIH)
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Cardiac Arrest; Cardiopulmonary Resuscitation
Keywords: CPR
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The design of this protocol is a prospective observational study to objectively measure the rate, depth and quality of chest compressions and ventilations delivered during cardiac arrest in the Pediatric Intensive Care Unit (PICU) and Emergency Department (ED) settings utilizing the MRx/Q-CPR. The data collected will be analyzed for several purposes - for comparison with current American Heart Association (AHA) Cardiopulmonary Resuscitation (CPR) guidelines and to determine chest wall stiffness for CPR modeling efforts and construction of biofidelic manikins or test dummies for CPR and auto safety.

DETAILED DESCRIPTION:
Context: Cardiopulmonary Resuscitation (CPR) guidelines recommend target values for selected CPR parameters related to rate and depth of chest compressions and ventilations, and avoidance of CPR-free intervals. Recent studies on adult patients however show that rescuers often do not adhere to these guidelines. There is currently very little data on the quality of CPR performed on pediatric patients, but given the close similarity in therapy it can be expected that the adherence to Guidelines is suboptimal for this patient group as well. Feedback on quality of chest compressions and ventilations delivered during CPR are most frequently guided by a subjective "code leader", and not objective measurements. Quantitative systems that provide CPR feedback have demonstrated improvement to adult patient treatment. Based on these studies, these feedback systems (termed Quality of CPR or Q-CPR systems) were further improved in a new device called Heartstart MRx with Q-CPR option (MRx/Q-CPR). These devices have been approved by the FDA for use for patients >8 years. The MRX/Q-CPR, attached by a cord to the defibrillator/monitor, detects, displays and records the rate, force and the depth of compressions through an accelerometer and force transducer inside the compression pad. These devices have currently been approved by the CHOP Resuscitation Committee and Medical device committee for clinical implementation in the CHOP Intensive Care units (ICU) and Emergency Department (ED).

Objectives: The goal of this study is to record and analyze the data from the MRx/Q-CPR during in-hospital cardiac arrests of children > 8 years for two research objectives. The primary research objective is to evaluate the rate, depth, and quality of chest compressions and ventilations delivered to children during in-hospital CPR. A secondary research objective is to determine the chest wall stiffness of children in order to improve quantitative CPR modeling efforts and to facilitate the construction of more biofidelic pediatric manikins for CPR simulation and test dummies for automotive safety

ELIGIBILITY:
Inclusion Criteria:

Cardiac Arrest Inclusion Criteria:

* Cardiac arrests occurring in the PICU or ED at The Children's Hospital of Philadelphia equipped with the MRx/Q-CPR
* Patient experiencing the arrest must be greater than or equal to 8 years old and receive chest compressions with the Q-CPR sensor employed

Clinical Staff Inclusion Criteria:

- All clinical staff who participate in resuscitation events in CHOP's ICU or ED

Exclusion Criteria:

* Cardiac arrests for patients classified as "do not attempt resuscitation" (DNAR) 1. CPR chest compressions without the Q-CPR device

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cardiac arrests occurring in the Pediatric Intensive Care Unit or Emergency Department at The Children's Hospital of Philadelphia equipped with the MRx/Q-CPR
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2006-06; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the rate, depth, and quality of chest compressions and ventilations delivered to children during in-hospital CPR. | Ongoing

SECONDARY OUTCOMES:
To determine the chest wall stiffness of children in order to improve quantitative CPR modeling efforts and to facilitate the construction of more biofidelic pediatric manikins for CPR simulation and test dummies for automotive safety. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Nadkarni, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States